CLINICAL TRIAL: NCT04082065
Title: Cyriax Manipulation in Lumbar Internal Derangement Syndrome
Brief Title: Cyriax Manipulation in Lumbar Derangement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahIU Sara yasin
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Derangement; Low Back
Keywords: Conventional physical therapy(CPT); .Low back pain (LBP),; Oswestery disability index (ODI),; Quality of life (QOL),; Range of motion (ROM); Visual analogue scale (VAS)
MeSH Terms: conditions — Low Back Pain; Hypotension

STUDY DESIGN:
Intervention Model Description: interventional
Who Masked: Investigator
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (Active Comparator): Myofacial release Stretching of hamstring and Piriformis
  Interventions: Other: conventional physical therapy
- cyriax lumber manipulation group (Experimental): Myofacial Release stretching of hamstrings and Piriformis Cyriax Lumbar Manipulation Techniques
  Interventions: Other: cyriax lumber manipulation group

INTERVENTIONS:
Other: conventional physical therapy — hot pack for 15 minutes Myofacial release (10 minutes) and Stretching of hamstrings and Piriformis (5 reps each with 2 second hold)
  Arms: conventional physical therapy
Other: cyriax lumber manipulation group — Hot Pack, Myofacial Release, stretching of hamstrings and Piriformis (five reps each with 2 seconds hold) and Cyriax Lumbar Manipulation Techniques
  Arms: cyriax lumber manipulation group

SUMMARY:
the objective of the study was to determine the effect of Cyriax manipulation for Pain, range of motion and quality of life in lumbar internal derangement radiculopathy in single physical therapy session. Randomized control trails were carried out in Railway general hospital from February 2018 to July 2018 in which 43 patients with Low back pain were randomly divided by lottery method into control and experimental group. Single session of treatment was given. tools used in the study are visual analog scale, Oswestry disability index and lumber range of motion. data was analysed through SPSS (statistical package for social sciences) 21.

DETAILED DESCRIPTION:
Human spine is a supporting structure of skeleton consisting of four curves cervical (lordosis), thoracic (kyphosis) , lumbar(lordosis) and sacrococcygeal (kyphosis). Cervical and lumbar being primary contributes for erect posture. Lumbar spine (lordotic curve) is the area of lower back of spine consisting of five vertebrae L1-L5 extending between thoracic and sacrum to accommodate progressively increasing loads.it is connected to pelvis where most weight bearing and body movement takes place. Over the last few decades, low-back pain has become increasingly problematic, placing significant burdens on economy and health system.the 2019 Global burden of Disease study estimated that low back pain is among the top ten diseases. low back pain is common that only a minority of individuals escape it. Eighty percent of anatomical and degenerative changes cause pain in lower back area .low back pain is extremely common having complex causes, may be acute sub-acute or chronic in nature depending upon severity of onset cause. Large forces acts on lumbar spine during functional activities such as lifting, running, walking and twisting causes repetitive micro traumas leading to low back pain which is distressing feelings.low back pain can be dull ache, shooting pain or burning sensation in nature originating from neuro-vascular, vertebral bones,facet joints or other vertebral structures. Low back pain which begin under 12th rib and on top of the inferior gluteal lines involving one or both lower extremities is called radiating low back pain which can be due to any internal derangement in anatomical structures of vertebral column. Internal derangement is disturbance of the regular order or arrangement of joint in which normal resting position of the articular surfaces of two adjacent vertebrae is disturbed as a result of a change in the position of fluid mechanics of disc, joint structure, ligaments, vascular and neuro-muscular system of lumbar spine due to mechanical or non mechanical stresses.Clinically lumbar internal derangement syndromes are .classified into mechanical and non mechanical based on origin internal derangement is disturbance of the regular order or arrangement of joint in which normal resting position of articular surfaces of two adjacent vertebrae is disturbed as a result of a change in position of fluid mechanics of disc, joint structures, ligaments, vascular and neuro-muscular system of lumbar spine due to mechanical or non mechanical stresses. Clinically lumbar internal derangement syndrome are classified into mechanical and non mechanical based on origin.Non mechanical internal derangement syndromes are due to non activity related disorders affecting spine such as inflammatory diseases (septic and hematological), tumors and infiltration lesions, metabolic disorders and acquired defects in neural arch whereas mechanical derangements are caused by placing abnormal stress on lower back disrupting normal order of lumbar spine anatomy. Physiotherapy treatments for low back pain includes myofascial release trigger point release, stretching of culprit muscles(hamstrings, lumbar erector spinae ,multifidus and piriformis), mobilization of vertebrae, traction of lumbar spine and Manipulation of lumbar spine (cyriax Manipulations, Osteopathic Manipulations and Chiropractor Manipulations).

Manipulations is passive movements carried out by clinician with single thrust high velocity, low amplitude or sustained pressure not under control of patient in order to return displacement to its proper position.Manipulations are used to reduce pain and disability caused by any internal derangement and intervertebral cartilaginous structure. Manipulations are based on different theories of which reduction of disc protrusions, correction of posterior joint dysfunction, mobilization of blocked vertebral joints and reduction of nerve root compression are some of them.

In 2012 John J Kuczynski conducted a systematic review on effectiveness of spinal manipulation therapy for treatment of chronic low back pain literature extracted from different data base concluded that spinal manipulations are safe and have significant clinical outcomes. A study published on 17th May 2018 on spinal manipulation in treatment of patient with MRI diagnosed lumbar disc herniation and sacroiliac hypermobility by Esmael Shokri et al concluded that lumbar and Sacro-iliac joint manipulations have significant effect on pain potential and disability. In March 2006 Muhammad A. Mohseni Bandpelet conducted randomized control trial study on spinal manipulation and ultrasound therapy in treatment of chronic low back pain. One hundred and twenty people were randomly allocated into manipulative group and ultrasound therapy group.They concluded that patient who received manipulative therapy showed greater decrease in pain intensity with increased spinal range of motions and functional qualities.

ELIGIBILITY:
Inclusion Criteria:

* lumber pain, pain radiating to leg, motor deficits in legs, , dural signs and symptoms, impaired nerve root mobility(straight leg raise and L3 stretch), back pain effecting Quality of life, ODI score less than 30 and Limited range of motion .

Exclusion Criteria:

* Osteoporosis of hip, Bilateral sciatica, having anticoagulant medication, pregnancy, patient with impaired mental status

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Owstery disability index | 3rd day
  ODI is self-reported tool used widely for measurement of functional disability related to. It was introduced by Fairbank et al in 1980 which gives guidelines for measuring functional disability due to LBP and considered gold standard. It is divided into 10 sections i.e. pain, personal care, sitting, walking, standing, travelling, weight lifting, sleeping, social life. Patient is guided to select one option according to their symptoms. Total score is 50.Once the individual score is calculated Percentage can be calculated by dividing it with total score i.e. 50 and then multiply it by 100.) In This study scores are calculated by filling the questionnaire before session and then filling it after two or three days after

SECONDARY OUTCOMES:
visual analog sclae | 1st day after session
  Visual Analogue Scale is an instrument used for measurement of characteristics that are in continuum manner and cannot be directly measured e.g. pain .it is simple and most widely used measurement for pain variations VAS is a horizontal line of 100 mm. Patient is asked to mark a point of their current status .it has 5-point description "nil" Mild'" moderate" "severe" and "very severe
range of motion lumber spine (flexion) | 1st day after session
  changes from baseline lumber flexion range of motion was taken by the help of goniometer
range of motion lumber spine (extension) | 1st day after session
  changes from baseline lumber range of motion was taken by the help of goniometer
range of motion lumber spine (right side bending) | 1st day after session
  changes from baseline lumber range of motion was taken by the help of goniometer
range of motion lumber spine (left side bending) | 1st day after session
  changes from baseline lumber range of motion was taken by the help of goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Scientific Group on the Burden of Musculoskeletal Conditions at the Start of the New Millennium. The burden of musculoskeletal conditions at the start of the new millennium. World Health Organ Tech Rep Ser. 2003;919:i-x, 1-218, back cover. PMID 14679827
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Punnett L, Pruss-Utun A, Nelson DI, Fingerhut MA, Leigh J, Tak S, Phillips S. Estimating the global burden of low back pain attributable to combined occupational exposures. Am J Ind Med. 2005 Dec;48(6):459-69. doi: 10.1002/ajim.20232. PMID 16299708
- [Background] Lidgren L. The bone and joint decade 2000-2010. Bull World Health Organ. 2003;81(9):629. Epub 2003 Nov 14. No abstract available. PMID 14710501
- [Background] Dionne CE, Dunn KM, Croft PR. Does back pain prevalence really decrease with increasing age? A systematic review. Age Ageing. 2006 May;35(3):229-34. doi: 10.1093/ageing/afj055. Epub 2006 Mar 17. PMID 16547119
- [Background] Ernst E, Canter PH. A systematic review of systematic reviews of spinal manipulation. J R Soc Med. 2006 Apr;99(4):192-6. doi: 10.1177/014107680609900418. PMID 16574972
- [Background] Ombregt L. A System of Orthopaedic Medicine-E-Book: Elsevier Health Sciences; 2013.
- [Background] Rubinstein SM, Terwee CB, Assendelft WJ, de Boer MR, van Tulder MW. Spinal manipulative therapy for acute low back pain: an update of the cochrane review. Spine (Phila Pa 1976). 2013 Feb 1;38(3):E158-77. doi: 10.1097/BRS.0b013e31827dd89d. PMID 23169072
- [Background] Assendelft WJ, Morton SC, Yu EI, Suttorp MJ, Shekelle PG. Spinal manipulative therapy for low back pain. A meta-analysis of effectiveness relative to other therapies. Ann Intern Med. 2003 Jun 3;138(11):871-81. doi: 10.7326/0003-4819-138-11-200306030-00008. PMID 12779297
- [Background] Aure OF, Nilsen JH, Vasseljen O. Manual therapy and exercise therapy in patients with chronic low back pain: a randomized, controlled trial with 1-year follow-up. Spine (Phila Pa 1976). 2003 Mar 15;28(6):525-31; discussion 531-2. doi: 10.1097/01.BRS.0000049921.04200.A6. PMID 12642755
- [Background] Wand BM, Bird C, McAuley JH, Dore CJ, MacDowell M, De Souza LH. Early intervention for the management of acute low back pain: a single-blind randomized controlled trial of biopsychosocial education, manual therapy, and exercise. Spine (Phila Pa 1976). 2004 Nov 1;29(21):2350-6. doi: 10.1097/01.brs.0000143619.34308.b4. PMID 15507794
- [Background] McMorland G, Suter E, Casha S, du Plessis SJ, Hurlbert RJ. Manipulation or microdiskectomy for sciatica? A prospective randomized clinical study. J Manipulative Physiol Ther. 2010 Oct;33(8):576-84. doi: 10.1016/j.jmpt.2010.08.013. PMID 21036279
- [Background] Muller R, Giles LG. Long-term follow-up of a randomized clinical trial assessing the efficacy of medication, acupuncture, and spinal manipulation for chronic mechanical spinal pain syndromes. J Manipulative Physiol Ther. 2005 Jan;28(1):3-11. doi: 10.1016/j.jmpt.2004.12.004. PMID 15726029
- [Background] Bialosky JE, Bishop MD, Robinson ME, Zeppieri G Jr, George SZ. Spinal manipulative therapy has an immediate effect on thermal pain sensitivity in people with low back pain: a randomized controlled trial. Phys Ther. 2009 Dec;89(12):1292-303. doi: 10.2522/ptj.20090058. Epub 2009 Oct 1. PMID 19797305